CLINICAL TRIAL: NCT04414371
Title: Tools for Wellbeing COVID-19 National Study of Undergraduate Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Tracy F. H. Chang, Ph.D., Associate Extension Specialist, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2020000953
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Stress; Anxiety; Depression; Resilience; Wellbeing; Mood
Keywords: yoga stress anxiety depression wellbeing COVID
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomized waitlist control cross over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Yoga Group (Experimental): Learn online yoga practices and practice daily for 12-weeks
  Interventions: Other: Yoga
- Group 2 - Control Group (Other): waist-list control for 4-week, cross-over to yoga practice for 8-week
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Yoga Namaskar and Nadi Shuddhi

SUMMARY:
The study evaluates the effectiveness of yoga practices on reducing stress, negative emotion, anxiety, and depression and on increasing positive emotion, wellbeing and resilience. The study uses randomized wait-list control. All U.S. undergraduate students in 4-year universities and colleges age 18 or older are eligible to participate.

DETAILED DESCRIPTION:
The purpose of this project is to widely disseminate a system of yoga tools to university students, faculty, and staff internationally to buffer the psychological impact of the COVID-19 pandemic. A recent study finds that stress, anxiety, and depression are the major psychological responses to COVID-19 during the early outbreaks in China (Wang et al., 2020). Globally, universities have closed campuses and moved learning, teaching, and working online with a very short notice. CDC suggests that keeping physically active and meditation are among the key activities to maintain a strong immune system and mental health during quarantine. Studies have documented physical and mental benefits of yoga practices (Balasubramaniam, Telles, & Doraiswamy, 2013; Brems, 2015; Brunner, Abramovitch, & Etherton, 2017; Büssing, Michalsen, Telles, Sherman, & Khalsa, 2012) This project introduces a system of yoga tools to buffer the psychological impact of COVID-19. This system of yoga tools is designed by Sadhguru Jaggi Vasudev, a yogi, mystic, author, and founder of the Isha Foundation. The Isha foundation is a volunteer-based international non-profit organization, offering yoga and meditation programs for human wellbeing and global harmony. In partnership with the Isha Foundation and Harvard University Medical School, the study will document the short-term and long-term effects of these yogic practices on stress, mood, wellbeing, resilience, and academic engagement for students and work engagement for faculty and staff during this challenging time.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Enrolled in 4-year universities/colleges in 2020
* Not graduate in May 2020

Exclusion Criteria:

* Younger than 18
* Not enrolled in 4-year universities/colleges in 2020
* Graduate in May 2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress | Change from baseline stress at 1-Month
  10-item Perceived Stress Scale (PSS), score 0-40, higher the score, higher stress
Stress | Change from baseline stress at 2-Month
  10-item Perceived Stress Scale (PSS), score 0-40, higher the score, higher stress
Stress | Change from baseline stress in 3-Month
  10-item Perceived Stress Scale (PSS), score 0-40, higher the score, higher stress
Wellbeing | Change from baseline wellbeing in 2-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing
Wellbeing | Change from baseline wellbeing in 4-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing
Wellbeing | Change from baseline wellbeing in 6-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing
Wellbeing | Change from baseline wellbeing in 8-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing
Wellbeing | Change from baseline wellbeing in 10-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing
Wellbeing | Change from baseline wellbeing in 12-week
  14-item Warwick-Edinburgh Wellbeing Scale (WEMWBS), score14-70, higher score higher wellbeing

SECONDARY OUTCOMES:
Anxiety | Change from baseline anxiety in 2-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Anxiety | Change from baseline anxiety in 4-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Anxiety | Change from baseline anxiety in 6-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Anxiety | Change from baseline anxiety in 8-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Anxiety | Change from baseline anxiety in 10-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Anxiety | Change from baseline anxiety in 12-week
  2-item PHQ-4, score 2-8, higher score higher anxiety
Depression | Change from baseline depression in 2-week
  2-item PHQ-4, score 2-8, higher score higher depression
Depression | Change from baseline depression in 4-week
  2-item PHQ-4, score 2-8, higher score higher depression
Depression | Change from baseline depression in 6-week
  2-item PHQ-4, score 2-8, higher score higher depression
Depression | Change from baseline depression in 8-week
  2-item PHQ-4, score 2-8, higher score higher depression
Depression | Change from baseline depression in 10-week
  2-item PHQ-4, score 2-8, higher score higher depression
Depression | Change from baseline depression in 12-week
  2-item PHQ-4, score 2-8, higher score higher depression
Resilience | Change from baseline resilience in 1-month
  6-item Brief Resilience Scale (BRS), score 6-30, higher score higher resilience
Resilience | Change from baseline resilience in 2-month
  6-item Brief Resilience Scale (BRS), score 6-30, higher score higher resilience
Resilience | Change from baseline resilience in 3-month
  6-item Brief Resilience Scale (BRS), score 6-30, higher score higher resilience
Positive Affect | Change from baseline positive affect in 2-week
  10-item Positive Affect Scale, score - 10 to 50, higher score more positive affect
Positive Affect | Change from baseline positive affect in 4-week
  10-item Positive Affect Scale, score - 10 to 50, higher score more positive affect
Positive Affect | Change from baseline positive affect in 6-week
  10-item Positive Affect Scale, score - 10 to 50, higher score more positive affect
Positive Affect | Change from baseline positive affect in 8-week
  10-item Positive Affect Scale, score - 10 to 50, higher score more positive affect
Positive Affect | Change from baseline positive affect in 10-week
  10-item Positive Affect Scale, score - 10 to 50, higher score more positive affect
Positive Affect | Change from baseline positive affect in 12-week
  10-item Positive Affect Scale, score - 10 to 50, higher score higher positive affect
Negative Affect | Change from baseline negative affect in 2-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect
Negative Affect | Change from baseline negative affect in 4-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect
Negative Affect | Change from baseline negative affect in 6-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect
Negative Affect | Change from baseline negative affect in 8-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect
Negative Affect | Change from baseline negative affect in 10-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect
Negative Affect | Change from baseline negative affect in 12-week
  10-item Negative Affect Scale, score - 10 to 50, higher score higher negative affect

CONTACTS AND LOCATIONS:
Overall Officials: Tracy F Chang, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasubramaniam M, Telles S, Doraiswamy PM. Yoga on our minds: a systematic review of yoga for neuropsychiatric disorders. Front Psychiatry. 2013 Jan 25;3:117. doi: 10.3389/fpsyt.2012.00117. eCollection 2012. PMID 23355825
- [Background] Brems C. A Yoga Stress Reduction Intervention for University Faculty, Staff, and Graduate Students. Int J Yoga Therap. 2015;25(1):61-77. doi: 10.17761/1531-2054-25.1.61. PMID 26667290
- [Background] Brunner D, Abramovitch A, Etherton J. A yoga program for cognitive enhancement. PLoS One. 2017 Aug 4;12(8):e0182366. doi: 10.1371/journal.pone.0182366. eCollection 2017. PMID 28783749
- [Background] Bussing A, Michalsen A, Khalsa SB, Telles S, Sherman KJ. Effects of yoga on mental and physical health: a short summary of reviews. Evid Based Complement Alternat Med. 2012;2012:165410. doi: 10.1155/2012/165410. Epub 2012 Sep 13. PMID 23008738
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Froeliger BE, Garland EL, Modlin LA, McClernon FJ. Neurocognitive correlates of the effects of yoga meditation practice on emotion and cognition: a pilot study. Front Integr Neurosci. 2012 Jul 26;6:48. doi: 10.3389/fnint.2012.00048. eCollection 2012. PMID 22855674
- [Background] Gard T, Noggle JJ, Park CL, Vago DR, Wilson A. Potential self-regulatory mechanisms of yoga for psychological health. Front Hum Neurosci. 2014 Sep 30;8:770. doi: 10.3389/fnhum.2014.00770. eCollection 2014. PMID 25368562
- [Background] Schmalzl L, Powers C, Henje Blom E. Neurophysiological and neurocognitive mechanisms underlying the effects of yoga-based practices: towards a comprehensive theoretical framework. Front Hum Neurosci. 2015 May 8;9:235. doi: 10.3389/fnhum.2015.00235. eCollection 2015. PMID 26005409
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789